CLINICAL TRIAL: NCT00701883
Title: Multicenter Randomized Double-Blind Placebo and Active Comparator Controlled Parallel-group, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of MBX-8025 in Moderately Obese Hyperlipidemic Patients With/Out Concomitant Atorvastatin"
Brief Title: Safety and Benefit of MBX-8025 With and Without Commonly Used Statins in Moderately Overweight Patients With High Cholesterol
Acronym: MBX-8025
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 70,961; M8025-20711
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-05

CONDITIONS: Hyperlipidemia
Keywords: Cholesterol; Hyperlipidemia; HDL; LDL; Triglycerides; Dyslipidemia
MeSH Terms: conditions — Hyperlipidemias; Dyslipidemias | interventions — (2-methyl-4-(5-methyl-2-(4-trifluoromethyl-phenyl)-2H-(1,2,3)triazol-4-ylmethylsulfanyl)phenoxy)acetic acid; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo/Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- MBX-8025 50 mg/Placebo (Experimental)
  Interventions: Drug: Placebo; Drug: MBX-8025
- MBX-8025 100 mg/Placebo (Experimental)
  Interventions: Drug: Placebo; Drug: MBX-8025
- Placebo/Atorvastatin 20 mg (Active Comparator)
  Interventions: Drug: Placebo; Drug: Atorvastatin
- MBX-8025 50 mg/Atorvastatin 20 mg (Experimental)
  Interventions: Drug: Atorvastatin; Drug: MBX-8025
- MBX-8025 100 mg/Atorvastatin 20 mg (Experimental)
  Interventions: Drug: Atorvastatin; Drug: MBX-8025

INTERVENTIONS:
Drug: Placebo — 2 capsules, once a day for 8 weeks
  Arms: MBX-8025 100 mg/Placebo; MBX-8025 50 mg/Placebo; Placebo/Atorvastatin 20 mg; Placebo/Placebo
Drug: MBX-8025 — 2 capsules, once daily for 8 weeks
  Arms: MBX-8025 50 mg/Placebo
Drug: MBX-8025 — 2 capsule, once daily for 8 weeks
  Arms: MBX-8025 100 mg/Placebo
Drug: Atorvastatin — 2 capsules, once daily for 8 weeks
  Arms: MBX-8025 100 mg/Atorvastatin 20 mg; MBX-8025 50 mg/Atorvastatin 20 mg; Placebo/Atorvastatin 20 mg
Drug: MBX-8025 — 2 capsules, once daily for 8 weeks
  Arms: MBX-8025 50 mg/Atorvastatin 20 mg
Drug: MBX-8025 — 2 capsules, once daily for 8 weeks
  Arms: MBX-8025 100 mg/Atorvastatin 20 mg

SUMMARY:
A Multicenter Randomized, Double-Blind, Placebo-Controlled Study to evaluate the efficacy, safety and tolerability of MBX-8025, a novel PPAR-d agonist to treat hyperlipidemia, insulin resistance and obesity in overweight, hyperlipidemic patients, both as monotherapy and in combination with Atorvastatin

Total participation for each patient is approximately 16-17 weeks, which may include up to a 2 week screening period, 5 week run-in period, 8 week treatment period, and 2 week follow-up. During the run-in period patients taking statins, statin combination or Zetia will undergo a 'washout'. All patients will be instructed to follow a weight-maintenance diet (i.e., their same diet prior to entering the study). They will be asked to defer initiating any weight loss diets or meaningful changes in their activity level until after they have completed the study. Once randomized into the double blind study, patients will visit the clinic every two weeks thereafter until the end of the study. At the end of the 8-week treatment phase, the double-blind study medication will be discontinued. Patients will attend a follow up visit two weeks after their final dose for safety evaluation.

DETAILED DESCRIPTION:
Total participation for each patient is approximately 16-17 weeks, which may include up to a 2 week screening period, 5 week run-in period, 8 week treatment period, and 2 week follow-up. During the run-in period patients taking statins, statin combination or Zetia will undergo a 'washout'. All patients will be instructed to follow a weight-maintenance diet (i.e., their same diet prior to entering the study). They will be asked to defer initiating any weight loss diets or meaningful changes in their activity level until after they have completed the study. Once randomized into the double blind study, patients will visit the clinic every two weeks thereafter until the end of the study. At the end of the 8-week treatment phase, the double-blind study medication will be discontinued. Patients will attend a follow up visit two weeks after their final dose for safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years
* Female patients must not be pregnant or breast-feeding
* Patients must be moderately overweight
* All patients must have abnormal cholesterol levels or a history of abnormal cholesterol levels as defined by the protocol.
* Patients taking medication to lower their cholesterol must be willing, in some cases, to discontinue their medications during the study Stable weight (a history of increasing or decreasing no more than 6.6 lbs [3 kg]) for at least 2 months prior to the study;

Exclusion Criteria

* Cancer or a history of a cancer within 5 years before screening, other than some skin cancers
* Patients planning elective surgery during the study
* Patients with a history of diabetes mellitus at study onset
* History of intolerance to, or adverse effect from atorvastatin
* History of weight loss due to stomach bypass or eating disorder
* All patients may not have had a stroke, TIA, an acute myocardial infarction, angina pectoris, coronary intervention procedure (including but not limited to angioplasty, stent placement, coronary revascularization) lower extremity bypass procedure, systemic or intracoronary fibrinolytic therapy) within 5 months of screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Lipid levels will be measured in patients with hyperlipidemia to assess the benefits of the investigational drug | 8 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Brian Roberts, M.D., Study Director — Gilead Sciences
Locations (28):
- United States (28):
  - Radiant Research, Birmingham, Alabama
  - Anasazi Internal Medicine Research, Phoenix, Arizona
  - Diabetes/Lipid Management and Research Center, Huntington Beach, California
  - Radiant Research, Santa Rosa, California
  - Clinical Research Consulting LLC, Milford, Connecticut
  - Genesis Research International, Indianapolis, Indiana
  - Midwest Institute for Clinical Research Inc., Indianapolis, Indiana
  - L-Marc Research Center, Louisville, Kentucky
  - Maine Research Associates, Auburn, Maine
  - Health Trends Research LLC, Baltimore, Maryland
  - Troy Internal Medicine Research, Troy, Michigan
  - Bridgewater Medical Group, Bridgewater, New Jersey
  - Clifton-Wallington Medical Group, Clifton, New Jersey
  - Rochester Clinical Research, Albuquerque, New Mexico
  - United Medical Associates P.C., Binghamton, New York
  - Rochester Clinical Research, Rochester, New York
  - Southgate Medical Group, West Seneca, New York
  - Great Lakes Medical Research, Westfield, New York
  - PharmQuest, Greensboro, North Carolina
  - Crescent Medical Research, Salisbury, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - PHA-Adult Medicine, Philadelphia, Pennsylvania
  - Radiant Research, Greer, South Carolina
  - Tricities Medical Research, Bristol, Tennessee
  - Holston Medical Group Clinical Research, Kingsport, Tennessee
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Diabetes and Glandular Disease Research, San Antonio, Texas
  - Walla Walla Clinic, Walla Walla, Washington

REFERENCES:
- [Derived] Choi YJ, Roberts BK, Wang X, Geaney JC, Naim S, Wojnoonski K, Karpf DB, Krauss RM. Effects of the PPAR-delta agonist MBX-8025 on atherogenic dyslipidemia. Atherosclerosis. 2012 Feb;220(2):470-6. doi: 10.1016/j.atherosclerosis.2011.10.029. Epub 2011 Nov 16. PMID 22169113
- [Derived] Bays HE, Schwartz S, Littlejohn T 3rd, Kerzner B, Krauss RM, Karpf DB, Choi YJ, Wang X, Naim S, Roberts BK. MBX-8025, a novel peroxisome proliferator receptor-delta agonist: lipid and other metabolic effects in dyslipidemic overweight patients treated with and without atorvastatin. J Clin Endocrinol Metab. 2011 Sep;96(9):2889-97. doi: 10.1210/jc.2011-1061. Epub 2011 Jul 13. PMID 21752880